CLINICAL TRIAL: NCT04073147
Title: Chemotherapy Free Treatment With Venetoclax and Obinutuzumab for Relapsed / Refractory Primary CNS Lymphoma Patients (VENOBI-CNS Study) - A Phase IB Study to Assess the Pharmacokinetics in the Cerebrospinal Fluid
Brief Title: Venetoclax and Obinutuzumab for Relapsed/Refractory Primary CNS Lymphoma
Acronym: VENOBI-CNS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Klinikum Stuttgart (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ML40029
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Primary CNS Lymphoma
Keywords: venetoclax; obinutuzumab; pharmacokinetics
MeSH Terms: interventions — venetoclax; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Three sequential dosing groups. Starting with dosing group 1 (5 patients), followed by dosing group 2 (5 patients) if no dose limiting toxicities occur during dosing group 1, and finally followed by dosing group 3 (5 patients) if no dose limiting toxicities occur in dosing group 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dosing group 1 (Experimental): Venetoclax 600mg + Obinutuzumab 1000mg
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab
- Dosing group 2 (Experimental): Venetoclax 800mg + Obinutuzumab 1000mg
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab
- Dosing group 3 (Experimental): Venetoclax 1000mg + Obinutuzumab 1000mg
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Venetoclax — Venetoclax per os
  Other Names: Venclyxto
Drug: Obinutuzumab — ObintuzumabIV
  Other Names: Gazyvaro

SUMMARY:
This is a phase IB study investigating the pharmacokinetics of the combination venetoclax and obinutuzumab in the cerebrospinal fluid of patient with relapsed primary CNS lymphoma.

DETAILED DESCRIPTION:
This is a phase IB study investigating the pharmacokinetics of the combination venetoclax and obinutuzumab in the cerebrospinal fluid of patient with relapsed primary CNS lymphoma. Three dosing groups of venetoclax (600mg, 800mg, and 1000mg) are planned; dosing of obinutuzumab will be 1000mg for each dosing group. 15 patients are planned being included from two centers in Germany.

ELIGIBILITY:
Inclusion criteria:

1. Age at inclusion ≥ 18 to 80 years, in case of ECOG 0 to 1 age up to 85 years
2. Eastern Cooperative Group performance status (ECOG) ≤ 3
3. Evaluable lymphoma manifestation in the CNS, either contrast-enhanced lesion in the brain parenchyma or measurable meningeal lesions.
4. Biopsy proven CD20 positive PCNSL at initial diagnosis or previous relapse/progression (re-biopsy at study inclusion is not mandatory for inclusion, but strongly recommended if time in remission is longer than 24 months).
5. At least one prior HD-MTX containing chemotherapy application (MTX dosed at ≥ 1 g/m2 body surface area) before progression or relapse.
6. Confirmed relapsed or refractory PCNSL according to the IPCG response criteria with the following definition: Evidence of disease recurrence following PR/CR or uCR or no radiological response (SD or PD) as per the IPCG criteria to prior chemotherapy regimen(s), at least one of them containing high-dose methotrexate.
7. Absolute neutrophil count (ANC) of at least 1'500/μl
8. Platelet count of at least 50'000/μl
9. Adequate liver (alanine aminotransferase [ALAT] and AST ≤ 3.0 x upper limit of normal [ULN] and total bilirubin ≤ 1.5 x ULN) and kidney function (estimated ≥ 30ml/min creatinine clearance according to Cockgroft-Gault formula)
10. Written informed consent
11. Recovery from toxicity from previous anti-lymphoma treatment to ≤ grade 2

Exclusion criteria:

1. Known allergy to venetoclax or other components of the formulation
2. Known allergy to obinutuzumab or other components of the formulation
3. Primary ocular lymphomas without brain parenchymal involvement
4. Lymphoma relapse outside the CNS; extra CNS relapse needs to be ruled out by body CT scans (neck till pelvis) or PET-CT scans.
5. Contraindications for lumbar puncture at the discretion of the clinical investigator
6. Prior exposure to obinutuzumab or venetoclax
7. Other additional anti-lymphoma treatment, e.g. chemotherapy or radiotherapy
8. Active hepatitis B or C
9. HIV seropositivity
10. Chronic use of immunosuppressive drugs, e.g. steroids for systemic autoimmune disease
11. Active infections requiring treatment
12. Other active malignancies (except non-melanoma skin cancer). Prior malignancies without evidence of disease for at least 5 years are allowed
13. Patient is pregnant or breastfeeding, or expecting to conceive or father children within one year of finishing venetoclax and 18 months for obinutuzumab.
14. Prior allogeneic haematopoietic stem cell or solid organ transplantation
15. Therapeutic intervention in setting of other former interventional clinical trial within 30 days before the first IMP administration in VENOBI study; simultaneous participation in registry and diagnostic studies or follow up of an interventional trial is allowed
16. Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial
17. Known or persistent abuse of medication, drugs or alcohol
18. Person who is in a relationship of dependence/employment with the sponsor or the investigator
19. Administration of moderate or strong CYP3A inhibitors or inducers within 1 week of initiation of venetoclax dosing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of venetoclax and obinutuzumab | day 3, 15, and 28
  Serum concentration and CSF concentration (μg/ml)

SECONDARY OUTCOMES:
Dose limiting toxicities | Within the first 6 weeks
  Defined by CTCAE (version 5.0)
Best lymphoma response achieved during induction | During induction (3 months)
  According to IPCG criteria
Progression-free survival 1 (PFS1) | Up to 15 months
  Time from the date of first dose until date of progression, relapse or death, whichever occurs first
Overall survival | Up to 15 months
  Time from the date of first dose until date of death
Progression-free survival 2 (PFS2) | Up to 12 months
  Time from the start of maintenance venetoclax treatment at week 12 until date of progression, relapse or death, whichever occurs first.
Mutational landscape of lymphoma | At baseline
  NGS test based on FoundationOne Heme® platform

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Illerhaus, Prof, Study Chair — Klinikum der Landeshauptstadt Stuttgart gKAö
Locations (1):
- Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will by made available on a data depository (e.g. https://datadryad.org/) after study completion and publication of results.
Supporting Information: Analytic Code
Time Frame: after study completion and publication of results.
Access Criteria: not decided yet